CLINICAL TRIAL: NCT06574256
Title: Investigation of the Effect of Online Nursing Education Given to Patients Diagnosed With Gynecological Cancer and Receiving Chemotherapy on Symptoms, Quality of Life and Patient Satisfaction
Brief Title: Investigation of the Effects of Online Education Application on Gynecological Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, yşegül Beyazpınar KAVAKLIOĞLU, principal investigator, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CelalBayarU-LEE-ABK-01
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Gynecological Cancer
Keywords: gynecological cancer; symptom management; telenursing; quality of life; chemotherapy

STUDY DESIGN:
Intervention Model Description: The universe of the study consisted of 114 women. The sample of the study consisted of 90 women. Inclusion Criteria for the Study Patients diagnosed with gynecological cancer and starting chemotherapy treatment for the first time in the hospital Speaking Turkish, having no communication problems Agreeing to participate in the study voluntarily Patients aged 18 and over Exclusion Criteria for the Study Illiterate Do not have a smart phone or computer Receiving radiotherapy together with chemotherapy Patients who do not know they have been diagnosed with cancer The intervention and control groups were randomized according to the literature; taking into account age group, education status, type and stage of gynecological cancer.
  When determining the intervention and control groups, patients who applied to the chemotherapy unit on Monday and Tuesday were included in the intervention group, and patients who applied on Wednesday and Thursday were included in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Patients in the intervention group will receive online nursing education and their quality of life and symptom complaints will be monitored by the nurse who provides education during three cycles of chemotherapy. At the end of the third cycle, patients' satisfaction with this education will be determined.
  Interventions: Other: Chemotherapy symptom Management Online Education
- control group (No Intervention): Patients in the control group will receive routine nursing care. Patients in the control group will be monitored for quality of life and symptom complaints during three cycles of chemotherapy.

INTERVENTIONS:
Other: Chemotherapy symptom Management Online Education — Randomization was achieved and data collection began. Patients were given the "Chemotherapy Symptom Management Education Booklet" and were informed that they would be contacted by phone.
  In the second and third stages of data collection, they were called by phone on the 7th day after receiving chemotherapy treatment. The symptoms experienced by the patient were evaluated with the N-SDS and the quality of life was evaluated with the EORTC QLQ-C30. Online nursing education videos were sent to the women in the intervention group regarding the symptoms they experienced. The practices they performed from the suggestions in the education videos and education booklets sent were recorded on the nurse follow-up form.
  In the fourth stage, the practices specified in the third stage were repeated on the 7th day after the third chemotherapy course, and at this stage, the satisfaction of the women in the intervention group with the online education was evaluated.
  Other Names: Chemotherapy symptom Management; nursing online education
  Arms: intervention group

SUMMARY:
The aim of the study was to examine the effect of online nursing education given to women diagnosed with gynecological cancer and receiving chemotherapy. It was conducted as a randomized controlled experimental study. The study examined the effect of online nursing education given to patients in the intervention group diagnosed with gynecological cancer and receiving chemotherapy on symptoms, quality of life and patient satisfaction. The control group received routine nursing care.

DETAILED DESCRIPTION:
This study examined the effect of online nursing education given to women diagnosed with gynecological cancer and receiving chemotherapy. This randomized controlled experimental study was conducted in a public hospital in Balıkesir province between December 1, 2021 and June 1, 2024. The study sample consisted of 90 women (intervention=45, control=45). Online nursing education was given to women in the intervention group receiving chemotherapy. Patients in the control group received routine nursing care. The study used the women's descriptive characteristics questionnaire, disease and treatment questionnaire, European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Nightingale Symptom Assessment Scale, nurse follow-up form and patient satisfaction questionnaire. Data were collected during three chemotherapy cycles in four phases.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with gynecological cancer and who have started chemotherapy treatment for the first time in the hospital,

having gynecological cancer

receiving chemotherapy

Speak Turkish, have no communication problems,

Accept voluntarily to participate in the study,

Patients who are 18 years of age or older

Exclusion Criteria:

* Illiterate Patients who do not have a smart phone or computer Patients who receive radiotherapy together with chemotherapy Patients who do not know they have been diagnosed with cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients diagnosed with gynecological cancer and receiving chemotherapy
Enrollment: 90 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
EORT QLQ-C30 | three monhts
  EORT QLQ-C30: It consists of three main dimensions and 30 questions, namely general well-being, functional difficulties and symptom control.
Nightingale symptom assessment scale | three monhts
  Nightingale symptom assessment scale: This scale, consisting of 38 items, has three sub-dimensions, namely physical, social and psychological well-being.

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, | three monhts
  EORT QLQ-C30: It consists of three main dimensions and 30 questions: general well-being, functional difficulties and symptom control. İThe first 28 questions are Likert-type. The other two questions are evaluated as 1: very bad and 7: excellent. Each subscale of the scale is scored between 0-100. High scores from the sub-dimension and general quality of life indicate that the quality of life is high, and high scores from the symptom scale indicate that the symptoms experienced are at a high level.
Nightingale Symptom Assessment Scale | three months
  Nightingale symptom assessment scale: This scale, consisting of 38 items, has three sub-dimensions: physical, social and psychological well-being. This is a Likert-type scale. The total sub-dimension score is calculated by adding the item scores in each sub-dimension and dividing by the number of items. 0-4 points are taken in each subscale of the scale. A high score indicates that the level of being affected by problems caused by the disease/treatment is high.
patient satisfaction | one months
  score average is taken.

CONTACTS AND LOCATIONS:
Overall Officials: ayşegül beyazpınar kavaklıoğlu, student, Principal Investigator — Celal Bayar University; emre yanıkkerem, prof.dr., Study Director — Celal Bayar University
Locations (1):
- CelalBayarU, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No